CLINICAL TRIAL: NCT02495337
Title: Tissue Collection for Gastro-esophageal Cancer Primary Cell Line Establishment
Brief Title: Tissue Collection Protocol for Gastroesophageal Cancers
Status: Recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 14-8514
Record Dates: First submitted 2015-05-27; First posted 2015-07-13 (Estimated); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Tissue Banks

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biopsy Samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- TIssue Collection: Only one arm will be used to collect tissue from Esophageal Adenocarcinoma
  Interventions: Other: Tissue Collection

INTERVENTIONS:
Other: Tissue Collection

SUMMARY:
This proposed collection of primary tumor cells lines will benefit esophageal cancer research within the University Health Network. This collection of gastro-esophageal tumor samples will be used to grow primary tumor cell lines, which will provide researchers with ready samples of various gastro-esophageal cancers. This will help to address the issue of access to these cell lines due to the limited number of patients with gastro-esophageal tumors, and high rates of contamination.

DETAILED DESCRIPTION:
Samples will be collected during surgery, EGD, or other biopsy. The surgeon will resect a sample for the research coordinator and/or fellow who will collect the sample and take it back to the lab for processing. Samples collected will be in excess of standard samples that are sent for pathology. The surgeon will make sure that excess samples will not affect pathological diagnosis. In addition samples may be purchased from the National Cancer Institute's Cooperative Human Tissue Network.

ELIGIBILITY:
Inclusion Criteria:

* Patients with esophagogastric cancer and/or GERD +/- Barrett's esophagus who will undergo surgery and/or EGD as standard of care.

Exclusion Criteria:

* Patients who are not well enough to undergo surgery or EGD as standard of care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with esophagogastric cancer and/or GERD +/- Barrett's esophagus who will undergo surgery and/or EGD as standard of care.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-05 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Effectively culture, proliferate, and store primary gastro-esophageal cell lines in order to create a bank of primary esophageal / gastric cancers for research purposes | Ongoing
  The primary objective of this study is to determine an effective way to culture, proliferate, and store primary gastro-esophageal cell lines in order to create a bank of primary esophageal / gastric cancers or GERD with/without Barrett's esophagus for research purposes, in addition we will be creating organoids.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Yeung, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network: Toronto General Hospital, Toronto, Ontario, Canada